CLINICAL TRIAL: NCT00947401
Title: The Practice of Fluid Management in the Post-anesthetic Care Unit (PACU) of Shaare Zedek Medical Center in Patients Undergoing Elective Surgery: an Observational Study
Brief Title: Fluid Management After Surgery in the Post-Anesthetic Care Unit (PACU)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Yaacov Gozal, MD, Dept. of Anesthesiology, Shaare Zedek Medical Center, Jerusalem, Israel
Other Study IDs: 1234567
Record Dates: First submitted 2009-07-26; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Surgery
Keywords: Surgery, elective; Fluids; Post Anesthesia Care Unit; PACU; Fluid management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective post surgery patients

SUMMARY:
The objective of the present study is to describe the current practice of postoperative fluid management in the Post Anesthesia Care Unit (PACU) of the Shaare Zedek Medical Center, Jerusalem, Israel.

DETAILED DESCRIPTION:
The aim of this study is to follow and present the current practice of fluid administration in the PACUof Shaare Zedek Medical Center for an extended period of time as a first step towards establishing guidelines for postoperative fluid management.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yrs
* elective surgery
* ASA I-III

Exclusion Criteria:

* massive intraoperative blood loss
* non elective surgery
* pregnant women
* stay in the PACU < 15 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age > 18 yrs) after elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yaacov Gozal, MD, Principal Investigator — Shaare Zedek Medical Center; Sarah Shapira, RN, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel